CLINICAL TRIAL: NCT03709914
Title: Phase 1, Non-comparative, Open-Label Study of Pharmacokinetics and Safety of a Single-Dose of ZTI-01 (Fosfomycin for Injection) in Pediatric Subjects (<12 Years of Age)
Brief Title: PK Study of Single-Dose ZTI-01 in Children (<12 Years of Age)
Acronym: Pediatric_PK
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nabriva Therapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: ZTI-01-100
Record Dates: First submitted 2018-10-10; First posted 2018-10-17 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Pediatric ALL
Keywords: Pediatric PK
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Fosfomycin; Injections

STUDY DESIGN:
Intervention Model Description: multiple-center, non-comparative, open-label, PK study
Masking Description: Subjects <12 years of age, are assigned by age to one of five age based cohorts. Study is open label and not masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- ZTI-01 Cohort 1 ≥ 6 to <12 years of age (Experimental): ZTI-01 (fosfomycin IV) 100 mg/kg (single dose) Subjects weighing within the 3rd to < 97th percentile for age
  Interventions: Drug: ZTI-01 100 mg/kg
- ZTI-01 Cohort 2 ≥ 2 to <6 years of age (Experimental): ZTI-01 (fosfomycin IV) 100 mg/kg (single dose) Subjects weighing within the 3rd to < 97th percentile for age
  Interventions: Drug: ZTI-01 100 mg/kg
- ZTI-01 Cohort 3a Birth to < 3 mos of age (Experimental): ZTI-01 (fosfomycin IV) 75 mg/kg (single dose) Subjects weighing within the 3rd to < 97th percentile for age
  Interventions: Drug: ZTI-01 75 mg/kg
- ZTI-01 Cohort 3b ≥ 3 to < 6 mos of age (Experimental): ZTI-01 (fosfomycin IV) 100 mg/kg (single dose) Subjects weighing within the 3rd to < 97th percentile for age
  Interventions: Drug: ZTI-01 100 mg/kg
- ZTI-01 Cohort 3c ≥ 6 to < 24 mos of age (Experimental): ZTI-01 (fosfomycin IV) 100 mg/kg (single dose) Subjects weighing within the 3rd to < 97th percentile for age
  Interventions: Drug: ZTI-01 100 mg/kg

INTERVENTIONS:
Drug: ZTI-01 100 mg/kg — ZTI-01 intravenous (IV)
  Other Names: IV fosfomycin; fosfomycin disodium; fosfomycin for injection
  Arms: ZTI-01 Cohort 1 ≥ 6 to <12 years of age; ZTI-01 Cohort 2 ≥ 2 to <6 years of age; ZTI-01 Cohort 3b ≥ 3 to < 6 mos of age; ZTI-01 Cohort 3c ≥ 6 to < 24 mos of age
Drug: ZTI-01 75 mg/kg — ZTI-01 intravenous (IV)
  Other Names: IV fosfomycin; fosfomycin disodium; fosfomycin for injection
  Arms: ZTI-01 Cohort 3a Birth to < 3 mos of age

SUMMARY:
Phase 1 study, a single dose of ZTI-01 given to pediatric subjects (under 12 years of age) who require antibiotic therapy to see what the body does to the drug (pharmacokinetics) and to compare if these effects are similar to those observed in adults at a 6g ZTI-01 dose. Study will help establish pediatric dosing in younger children by age cohort. This is a multiple-center, open-label, PK study of ZTI-01 (fosfomycin for injection) single dose scaled by allometric weight-modeling from an adult ZTI-01 dose of 6 grams. Eligible subjects must be receiving standard of care antibiotics for proven or suspected bacterial infection or for peri-operative prophylaxis surgery (in or out of hospital).

DETAILED DESCRIPTION:
Based on pre-dose weight on Day -1, subjects weighing within the 3rd to < 97th percentile based on age - will receive a single, weight adjusted dose of ZTI-01 via continuous IV infusion or syringe pump over a 1- hour (+10 min) period. Pediatric subjects participating in this study will be assigned to one of three cohorts based on age:

Cohort 1: ≥ 6 years to <12 years (n=6 PK evaluable subjects) Cohort 2: ≥ 2 years to <6 years (n=6 PK evaluable subjects)

Cohort 3: Birth to < 2 years (n=9 PK evaluable subjects), split into 3 subgroups:

(3a) Birth (defined as full term: 37 weeks of gestations or greater) to < 3 mos, (3b) ≥ 3 mos to < 6 mos, (3c) ≥ 6 mos to < 24 months

Cohorts 1 and 2 will be enrolled first with safety and PK data evaluated before enrolling the youngest Cohort 3. Blood for fosfomycin concentration measurement will be collected throughout the study. Safety will be assessed by monitoring adverse and serious adverse events based on medical history, vital signs, ECG, laboratory assessment and physical examination.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent/assent
* Male or female subjects aged from Birth (defined as full term: 37 weeks of gestation or greater) but less than 12 years old
* Hospitalized, currently receiving antibacterial treatment for confirmed or suspected bacterial infection
* If of reproductive potential, agrees to avoid becoming pregnant or impregnating a partner from the time of consent through 24 hours after completion of study drug administration
* Has sufficient intravascular access to receive study drug through peripheral or central line

Exclusion Criteria:

* Has history of known allergy, hypersensitivity, or intolerance to oral or intravenous fosfomycin
* Screening serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3x ULN or total bilirubin >2x ULN
* Female is post onset of menarche and currently pregnant, or breast feeding, or has a positive serum or urine β-human chorionic gonadotropin (β-hCG) pregnancy test
* Impaired renal function at screening based on the Revised Schwartz Formula using actual body height
* Known infection with immunodeficiency virus (HIV), hepatitis C virus, or hepatitis B virus
* Other laboratory tests, obtained as standard of care, that are outside the normal limits, considered by the Investigator, to be clinically significant
* Have surgery scheduled during collection period of plasma for fosfomycin concentrations
* Weighs outside of the 3rd to less than <97th percentile based on age
* History of a seizure disorder requiring ongoing treatment with anticonvulsive therapy or prior treatment with anti-convulsive therapy within the last 3 years
* Is currently participating in or has participated in an interventional clinical trial with an investigational compound or device within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) of administration of the study drug
* Has enrolled previously in the current trial or has received ZTI-01 or fosfomycin (IV or oral) for any other reason within the last 30 days
* Is expected to survive less than 72 hours after completion of study drug administration
* Plans to use cardiopulmonary bypass, extracorporeal membrane oxygenation, hemodialysis, or peritoneal dialysis during the study
* Clinically significant abnormalities on the ECG; or have or be at risk for major cardiac events or dysfunction including QTc prolongation, clinically unstable cardiac disease, receipt within 24 hours before the start of study drug of a medication that is labelled to prolong the QT interval, and for breastfed infant subjects only - receipt by the subject's mother within 24 hours before the start of study drug of a medication that is labelled to prolong the QT interval
* Planned blood transfusion within 24 hours of study drug administration or expected before the end of the PK sampling, or has had significant blood loss (≥5% of total blood volume) within 4 weeks before the screening visit
* Any condition that, in the opinion of the PI, would compromise the safety of the subject or the quality of the data
* Subject or caregiver/parent is unable or unwilling to adhere to the study-specified procedures and restrictions

Max Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Estimated)
Dates: Start 2018-05-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Area under plasma concentration-time curve (AUC) after a single dose of ZTI-01 | From time end of 1-hour infusion on Day 1, up to 8-12 hours post infusion on Day 1
  By age cohort, determine the ZTI-01 pharmacokinetic area under the plasma concentration-time curve

SECONDARY OUTCOMES:
Safety: Treatment Emergent Adverse Events (TEAE) | Baseline (start of dosing) through end of study follow-up (Day 2)
  Number and Incidence of TEAEs by age cohort
Maximum concentration (Cmax) after a single dose of ZTI-01 | From time end of 1-hour infusion on Day 1, up to 8-12 hours post infusion on Day 1
  By age cohort, determine the ZTI-01 pharmacokinetic maximum concentration (Cmax)

CONTACTS AND LOCATIONS:
Overall Officials: John S Bradley, MD, Principal Investigator — Rady Children's Hospital / Department of Pediatrics, University of California, School of Medicine; Jennifer Schranz, MD, Study Chair — Nabriva Therapeutics
Locations (5):
- United States (5):
  - Children's Hospital of Orange County, Orange, California
  - Rady Children's Hospital, San Diego, California
  - Kosair Charities Pediatric Clinical Research Unit, Louisville, Kentucky
  - Children's Hospital of Michigan, Detroit, Michigan
  - University of New Mexico Hospital, Albuquerque, New Mexico

IPD SHARING:
Plan to Share IPD: No